CLINICAL TRIAL: NCT00816361
Title: A Phase 1, Multicenter, Open-label, Single-arm, Dose-escalation Study to Evaluate the Safety, Tolerability, and Antitumor Activity of MEDI-573, a Fully Human Monoclonal Antibody Directed Against Insulin-like Growth Factors I and II, in Subjects With Advanced Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy Exists
Brief Title: A Dose-escalation Study to Evaluate the Safety, Tolerability, and Antitumor Activity of MEDI-573 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP184
Record Dates: First submitted 2008-12-23; First posted 2009-01-01 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — dusigitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- MEDI-573 0.5 mg/Kg QWk Dose Escalation (Experimental): Participants received MEDI-573 0.5 milligram per kilogram (mg/kg) as a 60-minute intravenous (IV) infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 1.5 mg/Kg QWk Dose Escalation (Experimental): Participants received MEDI-573 1.5 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 5 mg/Kg QWk Dose Escalation (Experimental): Participants received MEDI-573 5 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 10 mg/Kg QWk Dose Escalation (Experimental): Participants received MEDI-573 10 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 15 mg/Kg QWk Dose Escalation (Experimental): Participants received MEDI-573 15 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 30 mg/Kg Q3Wk Dose Escalation (Experimental): Participants received MEDI-573 30 mg/kg as a 90-minute IV infusion once every 21 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 45 mg/Kg Q3Wk Dose Escalation (Experimental): Participants received MEDI-573 45 mg/kg as a 90-minute IV infusion once every 21 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 5 mg/Kg QWk Dose Expansion (Experimental): Participants received MEDI-573 5 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573
- MEDI-573 15 mg/Kg QWk Dose Expansion (Experimental): Participants received MEDI-573 15 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
  Interventions: Drug: MEDI-573

INTERVENTIONS:
Drug: MEDI-573 — Administered at a dose determined by the subject's enrollment cohort as an IV infusion as part of a 21 day treatment cycle.

SUMMARY:
Evaluate the safety and tolerability of MEDI-573 in adult subjects with advanced solid tumors refractory to standard therapy or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor for which no curative or standard therapies exist.
* Karnofsky Performance Status ≥60.
* Adequate hematological function.
* Adequate organ function.
* Women of non-child-bearing potential (defined as being >1 year post-menopausal) or using effective contraception, e.g., use of oral contraceptives with an additional barrier method (since the investigational product may impair the effectiveness of oral contraceptives), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, or total abstinence, from the time the informed consent is signed through 30 days after the last dose of MEDI-573. Male subjects with partners of child-bearing potential must be surgically sterile or use contraceptive method as described above from the time of the initiation of MEDI-573 through 30 days after the last dose of MEDI-573.

Exclusion Criteria:

* No prior treatment within 4 weeks of study drug administration.
* No concurrent therapy for treatment of cancer.
* No uncontrolled diabetes.
* New York Heart Association Grade ≥ 2 congestive heart failure.
* History of myocardial infarction, unstable angina, transient ischemic attack or stroke within the previous 6 months prior to study entry.
* Documented brain metastasis.
* Pregnancy or lactation or plans to become pregnant while on study.
* Clinically significant abnormality on ECG.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-03-09 (Actual); Primary Completion 2012-09-11 (Actual); Study Completion 2012-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Perez, MD, MSc, Study Director — MedImmune LLC
Locations (6):
- United States (6):
  - Research Site, Scottsdale, Arizona
  - Research Site, Jacksonville, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Philadelphia, Pennsylvania

REFERENCES:
- See also: MEDI-573_CP-184_Protocol_Redacted_16Jul14 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=17&filename=MEDI-573_CP-184_Protocol_Redacted_16Jul14.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 43 participants ((23 participants in dose-escalation phase and 20 participants in dose-expansion phase) were entered in the study and received the study treatment.
Period: Overall Study
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Started | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 10 | 10
Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Not Completed | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 9 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Not completed — Death | 4 | 3 | 3 | 3 | 1 | 1 | 3 | 7 | 8
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who had received any MEDI-573 treatment.
Groups:
- MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion: Participants received MEDI-573 5 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
- MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion: Participants received MEDI-573 15 mg/kg as a 60-minute IV infusion once every 7 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
- TOTAL: Total of all reporting groups
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | TOTAL
Number analyzed (Participants) | 4 | 3 | 14 | 3 | 13 | 3 | 3 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (12.2) | 67.0 (8.7) | 64.5 (13.7) | 68.0 (13.2) | 61.2 (8.6) | 58.3 (18.5) | 65.7 (4.5) | 62.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 2 | 3 | 2 | 2 | 18
  Male | 0 | 2 | 10 | 1 | 10 | 1 | 1 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 14 | 3 | 12 | 3 | 3 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 4
  White | 4 | 3 | 14 | 3 | 10 | 3 | 2 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: AEs were any unfavorable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with the use of MEDI-573, whether or not considered related to MEDI-573. A SAE was any AE that resulted in: death; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; was life-threatening; was a congenital anomaly/birth defect in the offspring of a study participant; or was an important medical event that may not have resulted in death, threatened life, or required hospitalization and that, based on appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes above. TEAEs were defined as AEs present at baseline that worsened in intensity after administration of MEDI-573, or events absent at baseline that emerged after administration of MEDI-573, up to 30 days after the last dose.
Time Frame: From the start of study treatment through 30 days after the last dose of MEDI-573, up to 3.5 years
Population: The Safety Population included all participants who had received any MEDI-573 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 14 | 3 | 13 | 3 | 3
Participants
  TEAEs | 4 | 3 | 13 | 3 | 13 | 3 | 3
  Treatment emergent SAEs | 2 | 1 | 4 | 1 | 6 | 0 | 3

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Description: An abnormal laboratory finding that was judged by the investigator to be medically significant was reported as an AE. TEAEs were defined as events present at baseline that worsened in intensity after administration of MEDI-573, or events absent at baseline that emerged after administration of MEDI-573, for the period extending to 30 days after the last dose.
Time Frame: From the start of study treatment through 30 days after the last dose of MEDI-573, up to 3.5 years
Population: The Safety Population included all participants who had received any MEDI-573 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 14 | 3 | 13 | 3 | 3
Participants
  Anemia | 2 | 1 | 1 | 2 | 2 | 0 | 0
  Thrombocytopenia | 0 | 0 | 1 | 2 | 0 | 0 | 0
  Leukopenia | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Lymphopenia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Red blood cell count decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  White blood cell count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  White blood cell count increased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood alkaline phosphatase increased | 1 | 0 | 1 | 1 | 3 | 0 | 1
  Aspartate aminotransferase increased | 0 | 1 | 2 | 0 | 2 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 2 | 0 | 2 | 0 | 0
  Blood creatinine increased | 1 | 0 | 1 | 0 | 2 | 0 | 0
  Weight decreased | 0 | 0 | 1 | 0 | 2 | 1 | 0
  Blood insulin increased | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Blood creatine increased | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Blood growth hormone increased | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Blood lactate dehydrogenase increased | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Breath sounds abnormal | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cardiac enzymes increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Electrocardiogram QT prolonged | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Glomerular filtration rate decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Heart rate increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lipase increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Protein total increased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Weight increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hematuria | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Renal failure | 0 | 0 | 0 | 0 | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Vital Signs and Physical Findings Abnormalities Reported as TEAEs
Description: Vital signs and physical findings included parameters such as heart rate, blood pressure, temperature, and respiratory rate. TEAEs were defined as events present at baseline that worsened in intensity after administration of MEDI-573 or events absent at baseline that emerged after administration of MEDI-573, for the period extending to 30 days after the last dose.
Time Frame: From the start of study treatment through 30 days after the last dose of MEDI-573, up to 3.5 years
Population: The Safety Population included all participants who had received any MEDI-573 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 14 | 3 | 13 | 3 | 3
Participants
  Pyrexia | 1 | 1 | 1 | 0 | 1 | 0 | 0
  Tachycardia | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Breath sounds abnormal | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypotension | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Heart rate increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypertension | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Orthostatic hypotension | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Maximum Tolerated Dose (MTD) of MEDI-573
Description: The MTD was defined as the highest dose that can be safely administered to participants and was determined by the number of participants in each cohort with a dose-limiting toxicity (DLT). The number and proportion of participants in each dose cohort and the number of participants with a DLT was presented using the total number of participants in the MTD Evaluable Population as the denominator. 2 participants from Cohorts 0.5 and 5 mg/kg QWk (1 in each cohort) did not complete the DLT period and therefore not evaluable for MTD.
Time Frame: Cycle 1 Day 1 through Cycle 1 Day 21
Population: MTD Evaluable Population included all participants in dose-escalation phase who had received at least 1 full cycle of MEDI-573 and completed safety follow-up through DLT period (Cycle 1 Day 1 through Cycle 1 Day 21), or who experienced a DLT. Two participants did not receive a full cycle of MEDI-573 and therefore excluded from MTD population.
Measure: Number; unit: mg/kg
Groups:
- MEDI-573 Dose Escalation: Participants received MEDI-573 0.5 milligram per kilogram (mg/kg) up to 15 mg/kg as a 60-minute intravenous (IV) infusion once every 7 days or up to 45 mg/kg as a 90-minute IV infusion once every 21 days until unacceptable toxicity, documentation of disease progression, or other reason for participant withdrawal.
Arm/Group | MEDI-573 Dose Escalation
Number analyzed (Participants) | 21
mg/kg | NA — The MTD was not established in the study.

5. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any grade greater than or equal to (>=) 3 treatment-related non-hematologic toxicity that occurred during the DLT assessment period with the following exceptions: Grade less than (<) 4 serum-high glucose (fasting) with duration of < 24 hours; Grade 3 fever (in the absence of neutropenia) defined as > 40.0 degree centigrade (°C) [greater than (>) 104.0°F] that resolved to normal or baseline within 24 hours of treatment and was not considered an SAE; or Grade 3 rigors/chills that responded to optimal therapy; any Grade >= 3 treatment-related hematologic toxicity that occurred during the DLT assessment period.
Time Frame: Cycle 1 Day 1 through Cycle 1 Day 21
Population: The Safety Population included all participants who had received any MEDI-573 treatment.
Measure: Number; unit: Participants
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 14 | 3 | 13 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Optimal Biologically Effective Dose (OBED) of MEDI-573
Description: The OBED was defined as the dose at which all circulating insulin-like growth factor (IGF)-1 and IGF-2 ligand was sequestered by MEDI-573.
Time Frame: From the start of study treatment through 30 days after the last dose of MEDI-573, up to 3.5 years
Population: Safety population: Participants in the dose-escalation phase were analyzed for this outcome measure.
Measure: Number; unit: mg/kg
Arm/Group | MEDI-573 Dose Escalation
Number analyzed (Participants) | 23
mg/kg | 5

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) After the First Dose
Description: The Cmax was the maximum observed serum concentration of MEDI-573.
Time Frame: For weekly dosing: Pre- and post-infusion (0, 2, 6, 24, and 48 hours post-infusion); For 3 weekly dosing: Pre- and post-infusion (0, 2, 6, 24, and 48 hours post-infusion); and on Days 8 and 15
Population: The Safety Population included all participants who had received any MEDI-573 treatment. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 10 | 9
microgram per milliliter (mcg/mL) | 11.6 (5.54) | 71.8 (12.5) | 166 (37.7) | 264 (121) | 560 (251) | 588 (213) | 1200 (621) | 115 (42.6) | 412 (141)

8. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) After the First Dose
Description: The tmax was defined as actual sampling time to reach the maximum observed serum concentration of MEDI-573.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: Day
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 10 | 9
Day | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.06] | 0.04 [0.04 to 0.12] | 0.04 [0.04 to 0.14] | 0.28 [0.12 to 0.30] | 0.06 [0.06 to 0.06] | 0.06 [0.06 to 0.06] | 0.04 [0.04 to 0.30] | 0.06 [0.04 to 0.30]

9. Secondary Outcome: Trough Serum Concentration (Ctrough) After the First Dose
Description: The Ctrough was the lowest serum concentration of MEDI-573 within a dosing interval.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 9
mcg/mL | 1.04 (0.919) | 1.98 (0.377) | 17.3 (10.2) | 34.6 (26.8) | 138 (77.8) | 32.9 (28.2) | 63.5 (59.5) | 5.27 (4.80) | 77.8 (33.5)

10. Secondary Outcome: Dose Normalized Cmax (Cmax/Dose) After the First Dose
Description: The Cmax/dose was the dose-normalized maximum serum concentration of MEDI-573.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg/mL/mg
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 10 | 9
mcg/mL/mg | 0.319 (0.154) | 0.593 (0.122) | 0.401 (0.054) | 0.393 (0.129) | 0.422 (0.168) | 0.240 (0.072) | 0.352 (0.178) | 0.267 (0.110) | 0.314 (0.095)

11. Secondary Outcome: Area Under the Serum Concentration-time Curve Over the First Dosing Interval (AUCτ)
Description: Area under the serum concentration-time curve over the first dosing interval.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 9
mcg*day/mL | 9.59 (5.12) | 90.8 (18.6) | 431 (135) | 631 (288) | 1950 (917) | 3510 (1230) | 5790 (3390) | 227 (99.8) | 1280 (392)

12. Secondary Outcome: Dose-normalized Area Under the Serum Concentration Time Curve Over the First Dosing Interval (AUCτ/Dose)
Description: The AUCtau/dose was a measure of dose-normalized area under the serum concentration-time curve over the first dosing interval.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mcg*day/mL/mg
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 9
mcg*day/mL/mg | 0.245 (0.145) | 0.749 (0.176) | 0.962 (0.041) | 0.955 (0.401) | 1.47 (0.624) | 1.46 (0.526) | 1.70 (0.976) | 0.53 (0.233) | 0.981 (0.275)

13. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to MEDI-573
Description: Two methods were used to assess the immunogenicity data: an ECL-based method and measurement of neutralizing ADA. The titer was calculated by multiplying the minimum assay dilution factor by the reciprocal of the highest dilution factor which yielded an ECL multiple equal to or greater than the screening assay cut-point factor.
Time Frame: Pre-infusion on Day 1 of each cycle, end of treatment, and 90 days after last dose MEDI-573 (up to 3.5 years)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 10 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the proportion of participants with confirmed complete response (CR) or partial response (PR) according to the RECIST criteria The CR was defined as disappearance of all target and nontarget lesions and no new lesions; and PR was definded as >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline [screening]) and no new lesions.
Time Frame: From study entry through the end of the study, up to 3.5 years
Population: The Efficacy Evaluable Population included all participants who received MEDI-573 and had at least one tumor assessment after the initiation of treatment. Participants in the dose-expansion phase were to have at least 1 lesion that was measurable using RECIST criteria, and a histologically confirmed diagnosis of advanced urothelial carcinoma.
Measure: Number; unit: Percentage of Participants
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 13 | 3 | 12 | 3 | 1
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the duration from the start of treatment with MEDI-573 until the documentation of disease progression or death due to any cause, whichever occurred first.
Time Frame: From study entry through the end of the study, up to 3.5 years
Population: Efficacy Evaluable Population included all participants who received MEDI-573 and had at least 1 tumor assessment after initiation of treatment. Participants in dose-expansion phase had at least 1 measurable lesion and histologically diagnosis of advanced urothelial carcinoma. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 12 | 3 | 11 | 1 | 0
Months | 1.0 [0.5 to 1.5] | 2.6 [1.3 to 2.8] | 1.4 [1.2 to 2.8] | 1.5 [0.7 to 4.7] | 1.3 [0.7 to 4.2] | NA [1.2 to NA] — Median and upper limit of 95 % confidence interval was not applicable, as only 1 participant was evaluable. |

16. Secondary Outcome: Time to Progression
Description: Time to disease progression (TTP) was defined as the duration from the start of treatment with MEDI-573 until the documentation of disease progression.
Time Frame: From study entry through the end of the study, up to 3.5 years
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 12 | 3 | 11 | 1 | 0
Months | 1.0 [0.5 to 1.5] | 2.6 [1.3 to 2.8] | 1.4 [1.2 to 2.8] | 1.5 [0.7 to 4.7] | 1.3 [0.7 to 4.2] | NA [1.2 to NA] — Median and upper limit of 95 % confidence interval was not applicable, as only 1 participant was evaluable. |

17. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from the start of treatment with MEDI-573 until death.
Time Frame: From study entry through the end of the study, up to 3.5 years
Population: as for outcome 15
Measure: Median (Full Range); unit: Months
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 4 | 3 | 9 | 3 | 9 | 1 | 1
Months | 5.3 [2.1 to 8.7] | 13.6 [1.9 to 20.2] | 12.3 [1.4 to 37.3] | 2.5 [1.3 to 8.6] | 4.0 [1.1 to 33.0] | 7.9 [1.4 to 7.9] | 4.7 [4.7 to 4.7]

18. Secondary Outcome: Time to Response (TTR)
Description: Time to response was defined as the duration from the start of treatment with MEDI-573 to the first documentation of objective response (confirmed CR or PR) and was only assessed in participants who had achieved objective response.
Time Frame: From study entry through the end of the study, up to 3.5 years
Population: Participants in efficacy evaluable population and who achieved objective response were analyzed. As no participants achieved objective response in this study, number of participants analyzed for this outcome measure were zero.
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the duration from the first documentation of objective response (confirmed CR or PR) to the first documented disease progression.
Time Frame: From study entry through the end of the study, up to 3.5 years
Population: as for outcome 18
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Suppression Profiles of IGF-I and IGF-II Post-Administration of MEDI-573
Description: The suppression profiles of both IGF-1 and IGF-2 post administration of MEDI-573 in relation to time course of antibody concentrations in serum were evaluated during treatment.
Time Frame: From the start of study treatment through 30 days after the last dose of MEDI-573, up to 3.5 years
Population: The Safety Population included all participants who had received any MEDI-573 treatment. Here, "N" and "n" represent number of participants analyzed for this outcome measure and at specific time points, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Expansion | MEDI-573 15 mg/Kg QWk Dose Expansion
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 10 | 9
nanogram per milliliter (ng/ml)
  IGF-I at 0.000 | 4.014 (2.177) | 9.264 (7.401) | 4.655 (3.437) | 1.721 (2.710) | 1.440 (0.812) | 2.693 (2.855) | 1.925 (1.374) | 1.749 (0.643) | 2.099 (1.128)
  IGF-I at 0.042: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-I at 0.042 | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 0.063: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0
  IGF-I at 0.063 |  |  |  |  |  | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |
  IGF-I at 0.125: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-I at 0.125 | 0.252 (0.111) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 0.292: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 0 | 0 | 9 | 8
  IGF-I at 0.292 | 0.345 (0.227) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 1.000 | 2.088 (0.964) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | 0.215 (0.117) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 7.000: number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 10 | 9
  IGF-I at 7.000 |  |  |  | 0.223 (0.115) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | 0.641 (0.546) | 0.196 (0.078)
  IGF-I at 7.042: number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-I at 7.042 | 0.201 (0.087) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 14.000: number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-I at 14.000 |  |  |  | 0.232 (0.130) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |  | 0.360 (0.166) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 14.042: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-I at 14.042 | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-I at 21.000: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 3 | 3 | 10 | 8
  IGF-I at 21.000 |  |  |  | 0.334 (NA) — Standard deviation can not be calculated as only one participant evaluated. | NA (0.000) — Below the limit of quantitation (0.313 ng/mL). | 0.265 (0.189) | 0.241 (0.147) | 0.336 (0.177) | NA (0.000) — Below the limit of quantitation (0.313 ng/mL).
  IGF-II at 0.000 | 2.773 (0.320) | 2.984 (1.753) | 2.431 (0.139) | 1.879 (1.020) | 1.872 (0.862) | 2.780 (0.694) | 4.093 (1.039) | 2.689 (0.882) | 2.213 (0.752)
  IGF-II at 0.042: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-II at 0.042 | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 0.063: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0
  IGF-II at 0.063 |  |  |  |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) |  |
  IGF-II at 0.125: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-II at 0.125 | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL)
  IGF-II at 0.292: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 0 | 0 | 9 | 8
  IGF-II at 0.292 | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 1.000 | 1.060 (0.828) | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 7.000: number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 10 | 9
  IGF-II at 7.000 |  |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 7.042: number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-II at 7.042 | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 14.000: number analyzed (Participants) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-II at 14.000 |  |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 14.042: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 10 | 9
  IGF-II at 14.042 | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). |  |  | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).
  IGF-II at 21.000: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 3 | 3 | 10 | 8
  IGF-II at 21.000 |  |  |  | NA (NA) — Mean was below the limit of quantitation (0.626 ng/mL). Standard deviation can not be calculated as only one participant evaluated. | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL). | NA (0.000) — Below the limit of quantitation (0.626 ng/mL).

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after the last dose of study drug, up to 3.5 years
Arm/Group | MEDI-573 0.5 mg/Kg QWk Dose Escalation | MEDI-573 1.5 mg/Kg QWk Dose Escalation | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 10 mg/Kg QWk Dose Escalation | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion | MEDI-573 30 mg/Kg Q3Wk Dose Escalation | MEDI-573 45 mg/Kg Q3Wk Dose Escalation
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/3 | 10/14 | 3/3 | 9/13 | 1/3 | 3/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 4/14 | 1/3 | 6/13 | 0/3 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 13/14 | 3/3 | 13/13 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-573 0.5 mg/Kg QWk Dose Escalation (N=4) | MEDI-573 1.5 mg/Kg QWk Dose Escalation (N=3) | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion (N=14) | MEDI-573 10 mg/Kg QWk Dose Escalation (N=3) | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion (N=13) | MEDI-573 30 mg/Kg Q3Wk Dose Escalation (N=3) | MEDI-573 45 mg/Kg Q3Wk Dose Escalation (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-573 0.5 mg/Kg QWk Dose Escalation (N=4) | MEDI-573 1.5 mg/Kg QWk Dose Escalation (N=3) | MEDI-573 5 mg/Kg QWk Dose Escalation and Expansion (N=14) | MEDI-573 10 mg/Kg QWk Dose Escalation (N=3) | MEDI-573 15 mg/Kg QWk Dose Escalation and Expansion (N=13) | MEDI-573 30 mg/Kg Q3Wk Dose Escalation (N=3) | MEDI-573 45 mg/Kg Q3Wk Dose Escalation (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (5) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 6 (7) | 2 (3) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 2 (3) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 8 (10) | 1 (2) | 2 (3)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood growth hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (3) | 8 (9) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.